CLINICAL TRIAL: NCT05199727
Title: Comparison of the Efficacy and Safety of Low Intensity Extracorporeal Shock Wave Therapy Versus On-demand Tadalafil for Erectile Dysfunction
Brief Title: Shock Wave vs. On-demand Tadalafil for Erectile Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Hosam Kotb, Principal investigator, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5/2021UROL9
Record Dates: First submitted 2021-12-20; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Erectile Dysfunction
Keywords: Erectile dysfunction; Shock wave; Clinical trial
MeSH Terms: conditions — Erectile Dysfunction | interventions — Extracorporeal Shockwave Therapy; Tadalafil; Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shockwave group (Experimental): This group will receive 6 sessions (2 per week) with average 6,000 shocks per session with the PiezoWave2 unit
  Interventions: Device: LI-ESWT
- Medical Treatment Group (Active Comparator): This group will receive self-administered Tadalafil on-demand
  Interventions: Drug: Tadalafil 20Mg Oral Tablet

INTERVENTIONS:
Device: LI-ESWT — Low intenisty shockwave therapy newly used for treatment of erectile dysfunction by applying 6 sessions on 3 weeks (2 sessions /week)
  Other Names: Shockwave therapy
  Arms: Shockwave group
Drug: Tadalafil 20Mg Oral Tablet — Patients on this arm will allocate on on-demand tadalafil 20 mg for treatment of ED
  Arms: Medical Treatment Group

SUMMARY:
The objective of this study is to evaluate the effectiveness and safety of focused Li-ESWT on 25 participants complaining of ED compared to 25 participants complaining of ED on medical treatment on a prospective clinical trial for 12 weeks.

DETAILED DESCRIPTION:
Penile erection is a very complex process which requires a delicate and coordinated equilibrium among the neurological, vascular and the tissue compartments. It also includes arterial dilation, trabecular smooth muscle relaxation, and activation of the corporeal veno occlusive mechanism.Erectile dysfunction is defined as persistent inability to achieve or maintain the erection that is sufficient to permit satisfactory sexual intercours. It has a multifactorial pathogenesis, one of them is vasculogenic ED that occurs due to diseases such as diabetes mellitus, hypertension, hyperlipidemia, smoking, or vascular occlusive disease.

ED is also the most commonly treated sexual disorder and it affects approximately 20% of adult males over the age of 20. Nowadays, there are several treatment solutions for patients with ED, either non-invasive or invasive but the phosphodiesterase 5 inhibitors are still the first-line therapy for ED.

However, PDE5-Is effect is limited due to their inability to improve penile blood flow for a time period that is sufficient to allow optimal oxygenation and recovery of Cavernosal vasculature. Also, they cannot improve spontaneous erections. Moreover, several patients ranging from 40% to 50% will not respond to drug therapy even after optimization approaches such as treatment combinations have been implemented.

Also, it was proven that the effect of long-term daily use of PDE5-Is on endothelial function has induced a short-term improvement in erectile function but probably not a longstanding one.

Another option for ED patients is the use of intracavernosal injections which is considered the second line of treatment. Although PDE5-Is and intracavernosal injections are effective and safe vasodilating agents, they are unable to alter the underlying predominant pathology in patients with vasculogenic ED (eg, cavernosal artery insufficiency).

Other options include the use of intraurethral injections, or vacuum constrictive devices that could serve as salvage therapy for patients who failed to respond to PDE5-Is. If the previous options failed or not preferred by the patient, penile prosthesis implantation would be the last resort treatment for ED.

Many trials were done to find a new treatment modality that would provide a rehabilitative or curative effect for ED. This modality should affect the endothelial function and improve penile hemodynamics. One of these modalities was low-intensity extracorporeal shockwave therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male patients
* ED at least for 6 months
* vasculogenic ED
* from 25-60 years old

Exclusion Criteria:

* psychological patents
* neurological patients
* younger than 25 years old
* older than 60 years old

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Erectile function assessed by International Index of Erectile Function-5 | 3 months
  We will asessess erectile function using International Index of Erectile Function-5 (IIEF-5) where scores ≤6, severe; 8-16, moderate; 17-21, mild; and 22-25, none.

SECONDARY OUTCOMES:
Erection hardness score | 3 months
  We will assess the Erection Hardness Score (EHS) was based on self-estimated rigidity, categorized using a scale of 1- 4: (1) the penis is larger but not hard, (2) the penis is hard but not hard enough for penetration, (3) the penis is hard enough for penetration but not completely hard, and (4) the penis is completely hard and fully rigid for coitus

CONTACTS AND LOCATIONS:
Overall Officials: fouad zanaty, professor, Study Director — Menoufia University
Locations (1):
- Menoufia University, Cairo, Egypt

REFERENCES:
- [Background] Dong L, Chang D, Zhang X, Li J, Yang F, Tan K, Yang Y, Yong S, Yu X. Effect of Low-Intensity Extracorporeal Shock Wave on the Treatment of Erectile Dysfunction: A Systematic Review and Meta-Analysis. Am J Mens Health. 2019 Mar-Apr;13(2):1557988319846749. doi: 10.1177/1557988319846749. PMID 31027441
- [Background] Clavijo RI, Kohn TP, Kohn JR, Ramasamy R. Effects of Low-Intensity Extracorporeal Shockwave Therapy on Erectile Dysfunction: A Systematic Review and Meta-Analysis. J Sex Med. 2017 Jan;14(1):27-35. doi: 10.1016/j.jsxm.2016.11.001. Epub 2016 Dec 13. PMID 27986492
- [Background] Mo DS, Zhan XX, Shi HW, Cai HC, Meng J, Zhao J, Shang XJ. [Efficacy and safety of low-intensity extracorporeal shock wave therapy in the treatment of ED: A meta-analysis of randomized controlled trials]. Zhonghua Nan Ke Xue. 2019 Mar;25(3):257-264. Chinese. PMID 32216245